CLINICAL TRIAL: NCT05176639
Title: A Multiple Ascending Dose (MAD) Safety, Tolerability and Efficacy Study of Veligrotug (VRDN-001), a Humanized Monoclonal Antibody Directed Against the IGF-1 Receptor, in Normal Healthy Volunteers (NHV(s) and Subjects With Thyroid Eye Disease (TED)
Brief Title: A Safety, Tolerability and Efficacy Study of Veligrotug (VRDN 001) in Healthy Volunteers and Participants With Thyroid Eye Disease (TED) ( THRIVE )
Acronym: THRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VRDN-001-101
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Eye Disease
Keywords: Thyroid Eye Disease; Thyroid-Associated Ophthalmopathy; Dysthyroid Ophthalmopathy; Graves Eye Disease; Graves Orbitopathy; Myopathic Ophthalmopathy; Congestive Ophthalmopathy; Edematous Ophthalmopathy; Infiltrative Ophthalmopathy; Thyroid-Associated Orbitopathy; Graves Disease
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 3 Cohort (THRIVE) veligrotug (VRDN-001) (Experimental): Participants with TED will be randomized to either veligrotug (VRDN-001) 10mg/kg or placebo.
  Interventions: Drug: VRDN-001 Phase 3 Cohort (THRIVE)
- Phase 3 Cohort (THRIVE) VRDN-001 Placebo (Placebo Comparator): Participants with TED will be randomized to either veligrotug (VRDN-001) 10mg/kg or placebo.
  Interventions: Drug: VRDN-001 Placebo

INTERVENTIONS:
Drug: VRDN-001 Phase 3 Cohort (THRIVE) — 5 IV Infusions of veligrotug (VRDN-001) 10mg/kg
  Arms: Phase 3 Cohort (THRIVE) veligrotug (VRDN-001)
Drug: VRDN-001 Placebo — 5 IV Infusions of veligrotug (VRDN-001) placebo
  Arms: Phase 3 Cohort (THRIVE) VRDN-001 Placebo

SUMMARY:
The investigational drug, veligrotug (VRDN-001), is a monoclonal antibody that inhibits the activity of a cell surface receptor called insulin-like growth factor-1 receptor (IGF-1R). Inhibition of IGF-1R may help to reduce the inflammation and associated tissue swelling that occurs in patients with thyroid eye disease (TED). The primary objective of this clinical trial is to establish the safety, tolerability, and efficacy of veligrotug, and the pharmacokinetic (PK) and pharmacodynamic (PD) profiles of veligrotug in active TED patients who received 10 mg/kg.

ELIGIBILITY:
Key Inclusion Criteria for Active TED Participants (THRIVE):

* Must have moderate to severe active TED with documented evidence of ocular symptoms or signs that began within 15 months prior to screening
* Must have Clinical Activity Score (CAS) of ≥ 3 on the 7-item scale for the study eye
* Must agree to use highly effective contraception as specified in the protocol
* Female TED participants must have a negative serum pregnancy test at screening

Key Exclusion Criteria for Active TED Participants (THRIVE):

* Must not have received prior treatment with another anti-IGF-1R therapy or any investigational agent for TED
* Must not have used systemic corticosteroids or selenium within 2 weeks prior to Day 1
* Must not have received rituximab, tocilizumab or other immunosuppressive agents or any other therapy for TED within 8 weeks prior to Day 1
* Must not have received an investigational agent for any condition with 8 weeks prior to Day 1
* Must not have a pre-existing ophthalmic condition in the study eye that in the opinion of the Investigator would confound interpretation of the study results
* Must not have had previous orbital irradiation or surgery for TED in the study eye
* Must not have a history of inflammatory bowel disease
* Must not have a history of or screening audiometry assessment of clinically significant (as determined by investigator) ear pathology, relevant ear surgery, or hearing loss
* Female TED participants must not be pregnant or lactating

Note: Prior thyroidectomy, radioactive iodine (RAI) treatment, or orbital decompression surgery limited to bone only are NOT exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Proptosis Responder Rate | Week 15
  Proptosis Responder Rate in the study eye (i.e., reduction of proptosis of ≥ 2 mm from baseline [without a corresponding increase of ≥ 2 mm in the fellow eye] as measured by exophthalmometer)

SECONDARY OUTCOMES:
Change from baseline in proptosis in the study eye | Week 15
  Change from baseline in proptosis in the study eye as measured by exophthalmometer
Proptosis Responder Rate in the most proptotic eye | Week 15
  Proptosis Responder Rate in the most proptotic eye as measured by MRI/CT
Change from baseline in proptosis in the most proptotic eye | Week 15
  Change from baseline in proptosis in the most proptotic eye as measured by MRI/CT
Change from baseline in CAS | Week 15
  Change from baseline in Clinical Activity Score (CAS) in the study eye
Overall Responder Rate | Week 15
  Overall Responder Rate comprising Proptosis Responder Rate as measured by exophthalmometer and Clinical Activity Responder Rate in the study eye
Clinical Activity Responder Rate in the study eye | Week 15
  Clinical Activity Responder Rate in the study eye
Diplopia Responder Rate | Week 15
  Diplopia Responder Rate (i.e., reduction in Gorman Subjective Diplopia Score of ≥1 from baseline for participants with baseline Gorman Subjective Diplopia Score >0)
Diplopia Resolution Rate | Week 15
  Diplopia Resolution Rate (i.e., reduction in Gorman Subjective Diplopia Score to 0 from baseline for participants with baseline Gorman Subjective Diplopia Score >0)
Proportion of participants with a CAS score of zero or one in the study eye | Week 15
  Proportion of participants with a CAS of zero or one in the study eye

CONTACTS AND LOCATIONS:
Locations (53):
- United States (29):
  - University of Colorado - Department of Ophthalmology, Aurora, California
  - The Private Office of Raymond Douglas, Beverly Hills, California
  - USC Roski Eye Institute, Los Angeles, California
  - MACRO Trials, Inc., Los Angeles, California
  - Amy Patel Jain, MD, Newport Beach, California
  - Byers Eye Institute/Stanford University, Palo Alto, California
  - Senta Clinic, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Sina Medical Center, Homestead, Florida
  - Med-Care Research Inc., Miami, Florida
  - Edward Jenner Research Group Center LLC, Plantation, Florida
  - Sarasota Retina Institue, Sarasota, Florida
  - Vision Medical Research Inc., Orland Park, Illinois
  - University Health Diabetes, Endocrinology & Nephrology Center, Kansas City, Kansas
  - KU Medical Center, University of Kansas, Kansas City, Kansas
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Weymouth, Massachusetts
  - Fraser Eye Care Center, Fraser, Michigan
  - Kahana Oculoplastic & Orbital Surgery, Livonia, Michigan
  - University of Minnesota, Department of Ophthalmology and Visual Neurosciences, Minneapolis, Minnesota
  - Advanced Research International, LLC, Las Vegas, Nevada
  - Rutgers-New Jersey Medical School-Newark, Newark, New Jersey
  - New York Eye Ear Infirmary of Mount Sinai, New York, New York
  - Baylor College of Medicine (BCM)-Opthalmology, Houston, Texas
  - Neuro-Eye Clinical Trials, Houston, Texas
  - Neuro-Ophthalmology of Texas PLLC, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - West Virgina University Eye Insitute, Morgantown, West Virginia
- Australia (2):
  - Sydney Eye Hospital, Sydney
  - North Shore Eye Surgery, Sydney
- France (4):
  - CHU d'Angers, Angers
  - CH Nice, Nice
  - Centre Hospitalier National D'ophtalmologie, Paris
  - AP-HP- Hopital de la Pitie Salpetriere, Paris
- Germany (2):
  - Universitatsmedizin Gottingen, Göttingen
  - Johannes Gutenberg-University Medical Center, Mainz
- Poland (5):
  - NZOZ E-Vita, Bialystok
  - Specjakistyczny Osrodek Okulistyczny Oculomedica, Bydgoszcz
  - Santa Familia PTG Lodz, Lodz
  - Panstwowy Instytut Medycsny MSWiA, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Polikinika SP ZOZ, Wroclaw
- Spain (8):
  - Clinica Bonanova de Cirugia Ocular, Barcelona
  - Hospital Arruzafa, Córdoba
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Complexo Hospiralario Universitario de Santiago-Hospital Medico-Ciruxico de Conxo, Santiago
  - Hospital Universitatio Virgen De La Macarena, Servicio de Oftalmologia, Seville
  - Hospital Universitario Miguel Servet, Servicio de Paseo Isabel La Catdlica1, Zaragoza
- United Kingdom (3):
  - Northwick Park Hospital, London, United Kingdon
  - Western Eye Hospital Imperial College NHS trust, London, United Kingdon
  - Guy's and St. Thomas NHS Trust, London, United Kingdon

IPD SHARING:
Plan to Share IPD: No